CLINICAL TRIAL: NCT02371499
Title: Effect of Lactobacillus Casei dg (Enterolactis Plus®) in Patient With Irritable Bowel Syndrome: Multicenter, Randomized, Double-blind, Cross-over, Placebo Controlled, Pilot Study
Brief Title: Effect of Lactobacillus Casei DG (Enterolactis Plus®) in Patient With Irritable Bowel Syndrome: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PROBE-IBS/14
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Lactobacillus casei dg; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1st Arm (Experimental): Treatment with Lactobacillus casei DG (Enterolactis plus®)
  Interventions: Dietary Supplement: Lactobacillus casei DG
- 2nd Arm (Placebo Comparator): Treatment with equivalent product without bacteria (Enterolactis placebo)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei DG — the patients will receive 1 capsule of Lactobacillus casei DG (Enterolactis plus®) twice daily for 4 weeks
  Other Names: Enterolactis plus®
  Arms: 1st Arm
Dietary Supplement: Placebo — the patients will receive 1 capsule of product without bacteria (Enterolactis placebo) twice daily for 4 weeks
  Arms: 2nd Arm

SUMMARY:
The aim of the study is to collect data for the assessment of the Lactobacillus casei DG (Enterolactis plus®) effect on overall abdominal pain/discomfort, symptoms and gut microbiota composition in patients with Irritable Bowel Syndrome.

DETAILED DESCRIPTION:
The aim of the study is to collect data for the assessment of the Lactobacillus casei DG (Enterolactis plus®) effect on overall abdominal pain/discomfort, symptoms and gut microbiota composition in patients with Irritable Bowel Syndrome. The investigators suppose that, due to the immunomodulatory action of probiotics, overall abdominal pain/discomfort and symptoms will improve, fecal Immunoglobulin A levels will change, pro-inflammatory cytokine levels will decrease and the production of regulatory cytokines as Interleukin 10 will improve following consumption of Lactobacillus casei DG (Enterolactis plus®).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and ≤ 65 years.
* A positive diagnosis of Irritable Bowel Syndrome regardless of bowel habit (both males and females), according to Rome III criteria.
* Negative outcome of barium enema or left colonoscopy within the previous two years.
* Negative relevant additional screening or consultation whenever appropriate.
* Ability of conforming to the study protocol.

Exclusion Criteria:

* Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant on the basis of predefined values.
* Ascertained intestinal organic diseases, including ascertained celiac disease or inflammatory bowel diseases (Crohn's disease, ulcerative colitis, diverticular disease, infectious colitis, ischemic colitis, microscopic colitis).
* Previous major abdominal surgeries.
* Active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment are also acceptable).
* Untreated food intolerance such as ascertained or suspected lactose intolerance, as defined by anamnestic evaluation or, if appropriate, lactose breath test.
* Assumption of probiotics or topic and/or systemic antibiotic therapy during the last month.
* Systematical/frequent assumption of contact laxatives.
* Females of childbearing potential, in the absence of effective contraceptive methods.
* Pregnant women.
* Inability to conform with protocol.
* Treatment with any investigational drug within the previous 30 days.
* Recent history or suspicion of alcohol abuse or drug addiction.
* Previous participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Abdominal pain/discomfort as measured by 11-point Numerical Rating Scale | 1 day
  evaluation performed using a daily 11-point Numerical Rating Scale scale from "0" (none) to "10" (very severe) - (responders are defined as patients with ≥ 30% reduction in the weekly mean abdominal pain and/or discomfort score, versus mean value of run-in period, in at least 2 weeks out of the 4 weeks of the treatment period)
Irritable Bowel Syndrome degree-of-relief as measured by 7-point balanced ordinal scale | 1 week
  evaluation performed using weekly 7-point balanced ordinal scale, where "1"="completely relieved", "4"="unchanged" and "7"="as bad as I can imagine" - (responders are defined as patients reporting "completely relieved"=score 1 or "considerably relieved"=score 2 in at least 2 weeks out of the 4 weeks of the treatment period)
Stool frequency and consistency as assessed by Bristol Scale | 1 day
Microbiota of fecal sample as characterized by Ion Torrent Personal Genome Machine sequencing of 16S ribosomal RNA-based amplicons | 4 weeks
Overall satisfaction with treatment as measured by Visual Analogue Scale | 4 weeks
Quality of life as measured by Short-Form 12 Items Health Survey | 4 weeks
  evaluation performed using the validated Short-Form 12 Items Health Survey (SF-12) on a scale of 0 to 100
Anxiety and Depression as assessed by Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  evaluation performed using Hospital Anxiety and Depression Scale (HADS): seven items each for anxiety and depression, with a 4-point Likert scale (0-3) for each item providing a minimum score of 0 and a maximum score of 21 on each sub-scale
Consumption of rescue medication | 1 day
Secretory Immunoglobulin A and cytokines levels in fecal samples as measured by ELISA test. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giorvanni Barbara, MD, Principal Investigator — Policlinico S. Orsola-Malpighi - Azienda Ospedaliero-Universitaria di Bologna
Locations (5):
- Italy (5):
  - Policlinico S.Donato, San Donato, Milano
  - U.O. Gastroenterologia Universitaria, Pisa, Pisa
  - Azienda ULSS 1, Belluno
  - Azienda Ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - Policlinico Universitario Campus Biomedico, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Barbara G, Stanghellini V. Biomarkers in IBS: when will they replace symptoms for diagnosis and management? Gut. 2009 Dec;58(12):1571-5. doi: 10.1136/gut.2008.169672. No abstract available. PMID 19923339
- [Background] Cremon C, Carini G, De Giorgio R, Stanghellini V, Corinaldesi R, Barbara G. Intestinal dysbiosis in irritable bowel syndrome: etiological factor or epiphenomenon? Expert Rev Mol Diagn. 2010 May;10(4):389-93. doi: 10.1586/erm.10.33. PMID 20465494
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Rajilic-Stojanovic M, Biagi E, Heilig HG, Kajander K, Kekkonen RA, Tims S, de Vos WM. Global and deep molecular analysis of microbiota signatures in fecal samples from patients with irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1792-801. doi: 10.1053/j.gastro.2011.07.043. Epub 2011 Aug 5. PMID 21820992
- [Background] Jeffery IB, O'Toole PW, Ohman L, Claesson MJ, Deane J, Quigley EM, Simren M. An irritable bowel syndrome subtype defined by species-specific alterations in faecal microbiota. Gut. 2012 Jul;61(7):997-1006. doi: 10.1136/gutjnl-2011-301501. Epub 2011 Dec 16. PMID 22180058
- [Background] Moayyedi P, Ford AC, Talley NJ, Cremonini F, Foxx-Orenstein AE, Brandt LJ, Quigley EM. The efficacy of probiotics in the treatment of irritable bowel syndrome: a systematic review. Gut. 2010 Mar;59(3):325-32. doi: 10.1136/gut.2008.167270. Epub 2008 Dec 17. PMID 19091823
- [Background] Madsen K, Cornish A, Soper P, McKaigney C, Jijon H, Yachimec C, Doyle J, Jewell L, De Simone C. Probiotic bacteria enhance murine and human intestinal epithelial barrier function. Gastroenterology. 2001 Sep;121(3):580-91. doi: 10.1053/gast.2001.27224. PMID 11522742
- [Background] Eun CS, Kim YS, Han DS, Choi JH, Lee AR, Park YK. Lactobacillus casei prevents impaired barrier function in intestinal epithelial cells. APMIS. 2011 Jan;119(1):49-56. doi: 10.1111/j.1600-0463.2010.02691.x. Epub 2010 Oct 25. PMID 21143526
- [Background] Corinaldesi R, Stanghellini V, Cremon C, Gargano L, Cogliandro RF, De Giorgio R, Bartesaghi G, Canovi B, Barbara G. Effect of mesalazine on mucosal immune biomarkers in irritable bowel syndrome: a randomized controlled proof-of-concept study. Aliment Pharmacol Ther. 2009 Aug;30(3):245-52. doi: 10.1111/j.1365-2036.2009.04041.x. Epub 2009 May 12. PMID 19438846
- [Background] Quigley EM, Tack J, Chey WD, Rao SS, Fortea J, Falques M, Diaz C, Shiff SJ, Currie MG, Johnston JM. Randomised clinical trials: linaclotide phase 3 studies in IBS-C - a prespecified further analysis based on European Medicines Agency-specified endpoints. Aliment Pharmacol Ther. 2013 Jan;37(1):49-61. doi: 10.1111/apt.12123. Epub 2012 Nov 1. PMID 23116208
- [Derived] Cremon C, Guglielmetti S, Gargari G, Taverniti V, Castellazzi AM, Valsecchi C, Tagliacarne C, Fiore W, Bellini M, Bertani L, Gambaccini D, Cicala M, Germana B, Vecchi M, Pagano I, Barbaro MR, Bellacosa L, Stanghellini V, Barbara G. Effect of Lactobacillus paracasei CNCM I-1572 on symptoms, gut microbiota, short chain fatty acids, and immune activation in patients with irritable bowel syndrome: A pilot randomized clinical trial. United European Gastroenterol J. 2018 May;6(4):604-613. doi: 10.1177/2050640617736478. Epub 2017 Oct 8. PMID 29881616